CLINICAL TRIAL: NCT04144231
Title: Cognitive Behavioral Therapy for Insomnia (CBT-I) in Schizophrenia - A Randomized Controlled Clinical Trial (SLEEPINS)
Brief Title: Cognitive Behavioral Therapy for Insomnia (CBT-I) in Schizophrenia(SLEEPINS)
Acronym: SLEEPINS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Finnish Institute for Health and Welfare (Other Government); Finnish Institute of Occupational Health (Other)
Responsible Party: Principal Investigator, Tiina M. Paunio, Professor of Psychiatry and Vice Dean of Education / Department of Psychiatry, Faculty of Medicine, University of Helsinki, Research Professor / National Institute for Health and Welfare, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1129003, TYH2018219, 30000
Record Dates: First submitted 2019-10-24; First posted 2019-10-30 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Insomnia; Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment-as-usual (TAU) (No Intervention): Treatment-as-usual (TAU) delivered by psychiatrists and psychiatric nurses in HUS Psychiatry Outpatient Clinic for Psychosis. Participants who randomized to TAU -group, may receive medication for insomnia, but they will not received CBT-I. Treatment-as-usual is included in all intervention groups.
- Internet-Based Cognitive Behavioral Therapy for Insomnia (Experimental): TAU and Internet-Based Cognitive Behavioral Therapy for Insomnia (iCBT-I) with the support of a therapist, delivered by mobile application (HUS iCBT-I): There will be seven manualized sessions, conducted at intervals of either every one or two weeks.
  HUS iCBT-I, is based on the same theoretical model of insomnia as described in Morin 2003 and Edinger 2015- and involves the same interventions as ordinary CBT-I: a structured treatment focusing on education, behaviors and cognitions. iCBT-I consists of psychoeducation about sleep, sleep restriction therapy, stimulus control, relaxation techniques, and challenging beliefs and perception of sleep.
  During the therapy, the therapist monitors progress at least once a week, sends messages to the participant, and answers any treatment-related questions. The aim of the feedback is to comment on exercises, clarify intervention and motivate the patient to persist the in carrying out the treatment and the requested behavioral changes.
  Interventions: Behavioral: iCBT-I
- Cognitive Behavioral Group Therapy for Insomnia (Experimental): TAU and Cognitive Behavioral Group Therapy for Insomnia (GCBT-I): There will be six 90-minute manualized sessions, conducted at intervals of either one or two weeks. One booster session will be conducted one month after the treatment. Each group will have 4-8 people. The content of the CBT-I group is based on CBT for insomnia (as described above) and a previously published insomnia treatment manual for psychotic patients (Waters 2017).To ensuring the rights, safety and wellbeing of participants during the COVID-19 (Coronavirus) pandemic, we produce GCBT-I via internet.
  Interventions: Behavioral: GCBT-I

INTERVENTIONS:
Behavioral: iCBT-I — Internet-Based Cognitive Behavioral Therapy for Insomnia (ICBT-I) with the support of a therapist, delivered by mobile application (HUS iCBT-I)
  Arms: Internet-Based Cognitive Behavioral Therapy for Insomnia
Behavioral: GCBT-I — Cognitive Behavioral Group Therapy for Insomnia (GCBT-I)
  Arms: Cognitive Behavioral Group Therapy for Insomnia

SUMMARY:
Sleep problems are pervasive in people with schizophrenia. In our study, our goal is to determine whether we can alleviate sleep symptoms and improve quality of life and well-being in patients with major psychiatric disorders through cognitive behavioral therapy (CBT) delivered via the internet or in groups.

At the same time, the study provides information on factors that are commonly associated with sleep and well-being in patients. The intervention study is conducted as a Randomized Controlled Clinical Trial (RCT), in which subjects are randomized into three groups: 1) Treatment as usual (TAU), 2) TAU and Internet-based therapy for insomnia (ICBT-I), and 3) TAU and group therapy for insomnia (GCBT-I).

DETAILED DESCRIPTION:
Sleep is important for well-being. Lack of sleep and poor quality of sleep (Insomnia) are risk factors for psychiatric and somatic diseases such as depression, cardiovascular disease, diabetes and memory disorders and increases the risk of cognitive errors and accidents.

Psychiatric patients suffer from a wide variety of sleep disorders. Insomnia symptoms are known to increase the likelihood of later depression and even the use of disability pensions due to depression.

Various sleep disorders are also common in patients with schizophrenia. Previous studies on schizophrenia have reported-, symptoms of insomnia, especially the problem of falling asleep and poor sleep quality, circadian rhythm disruption, hypersomnolence and nightmares among the patients.

Cognitive behavioural therapy for insomnia (CBT-I) is an evidence-based treatment for insomnia. CBT-I can be implemented as an individual treatment, on a group basis or via the internet. There is evidence that CBT-I can also be used to treat a patient with a major psychiatric disorders, but randomized clinical trials (RCT) have rarely been published. Our research is based on the hypothesis that symptoms of insomnia in patients with schizophrenia can improved by CBT-I and, further, by improving patients' sleep quality their health and quality of life can also be improved.

The present study is designed to investigate the effect of two different treatment programs as compared to treatment as usual (TAU). The purpose of this study is to determine whether CBT-I can help relieve sleep symptoms and improve quality of life and well-being in patients with schizophrenia. At the same time, the study provides information on factors that are commonly associated with sleep and well-being in patients with major psychiatric disorders. The intervention study is conducted as an RCT, in which subjects are randomized into three groups: 1) Treatment as usual (TAU), 2) TAU and Internet-based therapy for insomnia (ICBT-I), and 3) TAU and group therapy for insomnia (GCBT-I).

The aim of this ongoing randomized controlled trial is to recruit 84 - 120 participants from Hospital District of Helsinki and Uusimaa (HUS) Psychiatry Outpatient Clinics for Psychosis, and they have previously participated in the nationwide SUPER Finland study (a study on genetic mechanisms of psychotic disorders and a part of the Stanley Global Neuropsychiatric Genomics Initiative). The study is performed on a cycle basis with a target of 12 to 24 patients per cycle, randomly assigned to three intervention groups.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, patients must meet the following criteria:

1. Have previously participated in the nationwide SUPER Finland study (www.superfinland.fi, a study on genetic mechanisms of psychotic disorders and a part of the Stanley Global Initiative) and have given permission for subsequent contact.
2. Be currently in psychiatric care at HUS
3. Be 18 years of age or older
4. Have a serious mental disorder (schizophrenia or schizoaffective disorder)
5. Have a stable medical condition
6. Have self-reported sleep problems: difficulty falling asleep, difficulty staying asleep, poor quality of sleep, or dissatisfaction with sleep
7. Have access to an electronic inquiry and treatment program and use of e-mail
8. Be able to participate in a sleep group if randomized.

Exclusion Criteria:

Exclusion criteria include:

1. ongoing cognitive-behavioral psychotherapy
2. diagnosed sleep disorder such as sleep apnea
3. insufficient Finnish language skills (insomnia interventions are produced in Finnish, so good Finnish language skills are required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-09-06 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index score (ISI) (Morin 2011) | baseline, 12, 24 and 36 weeks from the baseline
  A 7-item questionnaire used to assess insomnia severity with a score ranging between 0 to 28. Each questionnaire item addresses an aspect about sleep that is rated by the respondent on a 5-point scale (i.e., 0=no problem to 4=very severe problem).
Change in the health-related quality of life (HRQoL) instrument 15D score (Sintonen, 2001) | baseline, 12, 24 and 36 weeks from the baseline
  The 15D is a generic, comprehensive, 15-dimensional, standardized, self-administered measure of health-related quality of life (HRQoL) that can be used both as a profile and single index score measure. The maximum score is 1 (no problems on any dimension) and the minimum score is 0 (being dead).

SECONDARY OUTCOMES:
Self-reported subjective sleep quality collected through a digital smartphone app (AIDO Healthcare) | baseline to week 36
  1-2 times a week by emoji scale 1-5
Self-reported subjective fatigue collected through a digital smartphone app (AIDO Healthcare) | baseline to week 36
  1-2 times a week by emoji scale 1-5
Self-reported subjective mood collected through a digital smartphone app (AIDO Healthcare) | baseline to week 36
  1-2 times a week by emoji scale 1-5
Self-reported variables for sleep quantity and quality (adapted from Partinen 1996) | baseline, 12, 24 and 36 weeks from the baseline
  Questions about sleep quantity and quality
Self-reported variables for chronotype (Horne 1976) | baseline, 12, 24 and 36 weeks from the baseline
  Questions about chronotype (morningness-eveningness-)
Self-reported variables for dreaming and nightmares (adapted from Sandman 2015) | baseline, 12, 24 and 36 weeks from the baseline
  Questions about dreaming and nightmares
Self-reported variables for tiredness, fatigue, subjective memory, stress and recovery (Lundqvist 2016) | baseline, 12, 24 and 36 weeks from the baseline
  Questions about tiredness, fatigue, subjective memory, stress and recovery. Scale 1(very good) to 5(very poor).
Self-reported variables for functional ability (adapted from Tuomi 1998). | baseline, 12, 24 and 36 weeks from the baseline
  Questions about functional ability. Scale 0(very poor) to 10(very good).
Self-reported variables for symptoms of depression (Korenke 2001) | baseline, 12, 24 and 36 weeks from the baseline
  Questions about symptoms of depression. Scale 0(not at all) to 3 (Almost Always)
Self-reported variables for symptoms of psychosis (adapted from Haddoc 1999), | baseline, 12, 24 and 36 weeks from the baseline
  Questions about presence, severity, and characteristics of hallucinations, delusions, confused and disturbed thoughts and lack of insight and self-awareness.
Self-reported variables for lifestyle | baseline, 12, 24 and 36 weeks from the baseline
  Questions about exercise, usage of caffeine, alcohol, nicotine.
Subjective measures of Dysfunctional Beliefs and Attitudes about Sleep (DBAS-16) (Morin 2007) | baseline, 12, 24 and 36 weeks from the baseline
  DBAS-16 is a 16-item self reported questionnaire to measure people's beliefs and attitudes about their personal sleep situations. Items are ranked from 0, strongly disagree, to 10, strongly agree. Total score is mean of all questions, with a higher score representing more dysfunctional beliefs and attitude about sleep.
Self-reported Feedback Questionnaire | 12 weeks
  Participants experiences from the intervention including habits of practice of the new skills, experience of the effect of the intervention on sleep, mood and lifestyle, alliance with the therapist, the positive and negative effects of the treatment are questioned after the treatment period.
Objective information on sleep from Actigraphy (ACG) data | baseline (1 week) and week 12(1 week)
  The dataset from ACG includes Total Sleep Time (TST), Wake After Sleep Onset (WASO) Bed time, Get up time, Time in bed, Sleep efficiency (SE), Sleep Onset Latency (SOL), One minute immobility and Fragmentation index
Objective information on circadian rhythms from Actigraphy (ACG) data | baseline (1 week) and week 12(1 week)
  The dataset from ACG includes Cosine peak, Light/Dark ratio, Lowest 5 onset, Maximum 10 onset, RA, IV and IS
Subjective sleep diary tracking | baseline (1 week) and week 12(1 week)
  Each morning after waking participants completed the Sleep Diary during the ACG -monitoring period to provide a daily record of self-reported bedtime, get-up time, sleep duration, and daytime naps.
Objective information on activity from EMFIT Sleep Tracker data (Emfit Ltd) | baseline to week 13
  EMFIT device measures heart rate, breathing rate, movement activity every 4 seconds, sleep staging every 30 seconds, and heart rate variability every 3 minutes.
Objective information on recovery of the autonomic nervous system from EMFIT Sleep Tracker data (Emfit Ltd) | baseline to week 13
  EMFIT device measures heart rate, breathing rate, movement activity every 4 seconds, sleep staging every 30 seconds, and heart rate variability every 3 minutes.
Cognitive performance is measure with the psychomotor vigilance test (PVT) (Basner 2011) via a web-based interface | baseline, 12, 24 and 36 weeks from the baseline
  PVT is a sustained-attention, reaction-timed task that measures the speed with which subjects respond to a visual stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M. Paunio, M.D., Ph.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
Upon completion of the clinical trial, data will be made available upon reasonable request and by the review of ethics Committee of the Hospital District of Helsinki and Uusimaa, Finland

REFERENCES:
- [Background] Basner M, Dinges DF. Maximizing sensitivity of the psychomotor vigilance test (PVT) to sleep loss. Sleep. 2011 May 1;34(5):581-91. doi: 10.1093/sleep/34.5.581. PMID 21532951
- [Background] Edinger JD, Carney CE 2015. Overcoming Insomnia: A Cognitive-Behavioral Therapy Approach. Workbook.Oxford University Press 2015
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lundqvist A, Mäki-Opas T (eds.). Health 2011 Survey - Methods. Terveyden ja hyvinvoinnin laitos, Raportti 8/2016. Helsinki 2016
- [Background] Morin C, Espie C 2003. Insomnia: A clinical Guide to assessment and treatment. New York. Springer.
- [Background] Morin C. 2003. Treating insomnia with behavioral approaches: evidence for efficacy, effectiveness, and practicality. In M. P. Szupa, J.D. Kloss & D.F. Dinges (toim), Insomnia. Principles and Management, s. 73-82. Cambridge University press
- [Background] Morin CM, Vallieres A, Ivers H. Dysfunctional beliefs and attitudes about sleep (DBAS): validation of a brief version (DBAS-16). Sleep. 2007 Nov;30(11):1547-54. doi: 10.1093/sleep/30.11.1547. PMID 18041487
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Partinen M, Gislason T. Basic Nordic Sleep Questionnaire (BNSQ): a quantitated measure of subjective sleep complaints. J Sleep Res. 1995 Jun;4(S1):150-155. doi: 10.1111/j.1365-2869.1995.tb00205.x. PMID 10607192
- [Background] Sandman N, Valli K, Kronholm E, Revonsuo A, Laatikainen T, Paunio T. Nightmares: risk factors among the Finnish general adult population. Sleep. 2015 Apr 1;38(4):507-14. doi: 10.5665/sleep.4560. PMID 25325474
- [Background] Sintonen H. The 15D instrument of health-related quality of life: properties and applications. Ann Med. 2001 Jul;33(5):328-36. doi: 10.3109/07853890109002086. PMID 11491191
- [Background] Tuomi T Ilmarinen J, Jahkola A, Katajarinne l, Tulkki A (1998) Work ability index. Finnish Institute of Occupational Healht, Helsinki
- [Background] Waters F, Ree M ja Chiu V. Delivering CBT for Insomnia in Psychosis - A clinical guide. New York, Routledge, 2017
- [Derived] Tanskanen TE, Wegelius A, Harkonen T, Gummerus EM, Stenberg JH, Selinheimo SIK, Alakuijala A, Tenhunen M, Paajanen T, Jarnefelt H, Kajaste S, Blom K, Kieseppa T, Tuisku K, Paunio T. Cognitive behavioural therapy for insomnia (CBT-I) in schizophrenia and schizoaffective disorder: protocol for a randomised controlled trial. BMJ Open. 2024 Jun 12;14(6):e076129. doi: 10.1136/bmjopen-2023-076129. PMID 38866575
- See also: a study on genetic mechanisms of psychotic disorders and a part of the Stanley Global Initiative — http://www.superfinland.fi/